CLINICAL TRIAL: NCT01761591
Title: Acrobat Coronary Stent System Effectiveness European Study (European Multicenter Effectiveness Randomized Study of Svelte Medical Systems Acrobat Stent on a Wire Compared to Other BMS PCI in de Novo Coronary Lesions) ACES Trial
Brief Title: Acrobat Coronary Stent System Effectiveness European Study
Acronym: ACES
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty to identify eligible patients: 8 centers contributed 54 patients in 6 months.
Sponsor: Svelte Medical Systems Europe (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Svelte_13-002; ID RCB: 2012-A00670-43 (Other: ANSM)
Record Dates: First submitted 2012-12-12; First posted 2013-01-07 (Estimated); Last update posted 2014-08-26 (Estimated); Status verified 2014-08

CONDITIONS: Coronary Artery Disease
Keywords: CAD; PCI; BMS; Svelte; Acrobat; direct stenting; RCT
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acrobat (Experimental): Device: PCI with Svelte Acrobat
  Interventions: Device: PCI with Svelte Acrobat
- Control BMS (Active Comparator): Device: PCI with other BMS
  Interventions: Device: PCI with other BMS

INTERVENTIONS:
Device: PCI with Svelte Acrobat — Percutaneous coronary intervention with Svelte Acrobat Coronary Stent System
  Arms: Acrobat
Device: PCI with other BMS — Percutaneous coronary intervention with any other routine use CE marked bare metal stent (BMS) implantable either via direct stenting or after lesion pre-dilation
  Arms: Control BMS

SUMMARY:
The purpose of this randomized controlled trial (RCT) is to demonstrate the clinical benefit and impact on resource utilization of percutaneous coronary interventions (PCI) with the Svelte Acrobat Stent System compared to any other CE marked bare metal stent (BMS) implantable via direct stenting or after lesion pre-dilation, in patients with coronary lesions that are eligible for direct stenting and who are recruited and treated so as to reflect real-life routine practice.

DETAILED DESCRIPTION:
The main objectives of this study are to test the following hypotheses:

1. The evaluated stent is clinically non-inferior to control BMS in terms of freedom of MACE
2. The evaluated stent is clinically beneficial compared to control BMS by reducing exposure to radiations, amount of contrast medium administered, procedure time, as well as amount of administered heparin,
3. The evaluated stent does not result in more frequent adverse events than control BMS,
4. The evaluated stent improves direct stenting success while not decreasing procedural success compared to control BMS.
5. Resource utilization (R.U.):

   1. Hospital-perspective resource utilization during the index admission and index procedure is not greater with evaluated the stent and potentially lower than with control BMS
   2. Resource utilization over a 6-month time-horizon, in relation to routine follow-up and MACE, is not greater with the evaluated stent than with control BMS.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for PCI and demonstrating native vessel or vein/arterial graft disease
* symptomatic CAD: either stable angina pectoris (CCS 1, 2, 3 pr 4) or unstable (Braunwald Class 1-3, B-C) or positive functional ischemia study
* Male and post-menopausal female
* Patient provides written informed consent prior to procedure
* Patient willing to comply with protocol
* Acceptable candidate for CABG
* Patient indicated for stenting of one or more de novo stenotic lesions in native coronary arteries or bypass grafts with or without direct stenting
* All target lesions for stenting in single or multi-vessel disease meet all inclusion criteria
* None of the lesions requires stenting with Drug eluting stents
* At least one lesion is visually estimated to be candidate for direct stenting
* All target lesions for stenting have a visually estimatd RVD >= 2.5 mm and <= 3.5 mm
* All target lesions for stenting are visually estimated to have LL =< 20 mm (to cover the lesion with 1 stent)
* All target lesions for stenting visually estimated to have a stenosis > 50% and < 99%
* All target lesions for stenting are ACS lesions TIMI flow >= 1

Exclusion Criteria:

* Currently enrolled in another clinical trial that has not completed the primary endpoint or that clinically interferes with the current study endpoints
* A previous coronary procedure within 30 days
* Any of the target lesion(s) requires treatment with a device other than PTCA prior to stent placement (such as, but not limited to, directional coronary atherectomy, excimer laser, rotational atherectomy, etc.)
* Previous BMS deployment anywhere in the target vessel within the past 6 months
* Any DES deployment anywhere in the target vessel within the past 9 months
* Any previous stent placement within 10 mm (proximal or distal) of the target lesion
* Patient has diabetes mellitus
* Co-morbid condition(s) that could limit the patient's participation or impact the trial
* Documented LVEF < 30% at the most recent evaluation
* Evidence of AMI within 72 hours of the intended trial procedure and/or with TIMI flow 0
* History of CVA or TIA in the last 6 months
* Leukopenia (<3.5 x 10^9/L)
* Neutropenia (<1000/mm3) <= 3 days prior to enrollment
* Thrombocytopenia (<10^5/mm3) pre-procedure
* Active peptic ulcer or active GI bleeding
* History of bleeding diathesis or coagulopathy or inability to accept blood transfusions
* Known hypersensitivity or contraindication to aspirin, heparin or bivalirudin, clopidogrel or ticlopidine, cobalt, nickel, L-605 Cobalt chromium alloy or sensitivity to contrast media, which cannot be adequately pre-medicated
* Serum creatinine level > 2.5 mg per dl within 7 days prior to index procedure
* In-stent restenosis
* Patient not able to give consent or read or write or protected by law or under guardianship or deprived of civil rights
* Woman of childbearing age
* Patient not covered by health or social insurance
* Unprotected left main CAD with obstruction > 50% , not protected by at least one non-obstructed bypass graft to the LAD or left circumflex (LCX) artery or their branches
* Target vessel exhibiting multiple lesions > 40% diameter stenosis outside of a range of 5 mm proximal and distal to the target lesion(s) to be stented based on visual estimate or on-line QCA
* Any target lesion for stenting exhibits an intraluminal thrombus (occupying > 50% of the true lumen diameter) at any time
* Any target lesion for stenting is excessively tortuous (two bends > 90° to reach the target lesion)
* Lesion location that is aorto-ostial or within 5 mm of the origin of the LAD or LCX
* Any target lesion for stenting is has side branches > 2.0 mm in diameter in which bifurcation stenting is planned
* Any target lesion >20 mm
* Any target lesion totally occluded (CTO)
* Any target lesion has TIMI flow = 0
* Any target lesion with ISR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients free of Major Adverse Cardiac Event ("MACE-free patients") | From the date and time of randomization until 6 months after the index procedure
  Major Adverse Cardiac Event ("MACE") is defined here as device-oriented composite endpoint that includes, in hierarchical order: Cardiac death (All deaths are considered cardiac unless an unequivocal non-cardiac cause can be established), Myocardial Infarction ("MI"), Target Lesion Revascularization ("TLR").

SECONDARY OUTCOMES:
administered dye | intra-procedural
  Volume (ml) of administered dye i.e. injected radiological contrast medium.
procedure duration | intra-procedural
  Procedure duration (minutes) from arterial access to closure.
radiation exposure | intra-procedural
  Radiation exposure (gY/cm²) & total fluoroscopy time (min)
acute success | procedure to discharge
  Acute success is measured at procedure end according to 4 criteria:
  1. Lesion success: Residual stenosis of the target lesion < 30% of the RVD using any percutaneous method.
  2. Direct stenting success: Lesion success without unplanned pre-dilation performed (planned pre-dilation is an exclusion criterion) from the trial.
  3. Device Success: Direct stenting success without post-dilatation or with post-dilatation using the Stent Delivery System (SDS).
  4. Procedure success: Lesion success & no in-hospital MACE
heparin administration | intra-procedural
  Amount of heparin administered during the procedure
adverse events | 6 months
  Adverse events occurrence:
  1. Death
  2. MI
  3. Repeat coronary revascularization
  4. Bleeding or vascular complications at discharge
  5. Stent thrombosis up to 6 months
  6. Other serious adverse events

OTHER OUTCOMES:
resource utilization | 6 months
  Resource utilization (R.U.) endpoints:
  Overall procedural and follow-up R.U. including:
  * Man-time
  * Facility usage
  * Amount of medical devices and drugs used:
    1. during index procedure
    2. after index procedure until discharge
    3. between discharge and 6-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jean Fajadet, MD, Principal Investigator — Clinique Pasteur, 45 avenue Lombez, Toulouse 31300, France, Tel. 33 (0)5 62 21 16 99 - secretariat@interv-cardio-toul.com; Andrew Schut, Study Director — Svelte Medical Systems, Inc., 675 Central Avenue, New Providence, NJ 07974, USA, Tel. 1.908.264.2181 - aschut@sveltemedical.com
Locations (12):
- Belgium (4):
  - OLV Ziekenhuis, Aalst
  - ZNA Middelheim - Hartcentrum, Antwerp
  - ZOL Sint Jan, Genk
  - CHU Liège - Sart Tilman, Liège
- France (7):
  - CHU Nord Grenoble - A. Michalon, La Tronche
  - AP-HP Hôpital Européen Georges Pompidou, Paris
  - AP-HP La Pitié Salpétrière, Paris
  - CHU Bordeaux Sud - Hôpital Cardiologique Haut Lévêque, Pessac
  - Clinique St Hilaire, Rouen
  - CHU Rangueil, Toulouse
  - Clinique Pasteur, Toulouse
- Hospital Universitari Vall d'Hebrón, Barcelona, Spain

REFERENCES:
- [Background] Piscione F, Piccolo R, Cassese S, Galasso G, D'Andrea C, De Rosa R, Chiariello M. Is direct stenting superior to stenting with predilation in patients treated with percutaneous coronary intervention? Results from a meta-analysis of 24 randomised controlled trials. Heart. 2010 Apr;96(8):588-94. doi: 10.1136/hrt.2009.183277. PMID 20357387
- [Background] Shao C, Stella PR, Agostoni P. Complex made easy: left anterior descending artery trifurcation lesion completely treated with a single device. J Invasive Cardiol. 2012 Aug;24(8):E164-6. PMID 22865317
- [Background] de Ribamar Costa J, Abizaid A, Stella P, Fernandez A, Granada J, Feres F, Serruys P. Preliminary results of the svelte trial: first-in-man assessment of the novel acrobat™ SOAW (Stent-On-A-Wire) coronary system. J Am Coll Cardiol. 2011;57(14s1):E1658-E1658. doi:10.1016/S0735-1097(11)61658-6